CLINICAL TRIAL: NCT06462534
Title: The Band-Frail Study: A Provincial Intervention to Outweigh Diabetes and Frailty in New Brunswick
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Martin Senechal, Full Professor, Martin Senechal, Ph.D., University of New Brunswick
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-029
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes; Frailty
Keywords: elastic band resistance training; exercise intervention; aging; community intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Band-Frail Intervention (Experimental): Individuals 65 years or older living with T2D and frailty will participate in elastic band resistance training and diabetes education sessions.
  Interventions: Behavioral: Band-Frail Program

INTERVENTIONS:
Behavioral: Band-Frail Program — Participants will complete 16 weeks of elastic band resistance training and diabetes management education.
  Exercise Component:
  The elastic band resistance training involves 12 exercises: chair sit-to-stands, seated chest press, seater upper back reverse fly, seated single arm row, seated single arm lateral raise, seated single arm bicep curl, seated single arm triceps extension, seated single leg quadriceps extension, standing hamstring curl, standing leg extension, and seated abdominal crunches.
  There will be a one-minute rest between each set and a self-determined rest period between exercises.
  Education Component:
  A certified Diabetes Educator and registered dietitian will present information to participants covering topics relating to T2D management and nutritional information.

SUMMARY:
The goal of this study is to test whether psychological, social, and physical health outcomes of older adults living with type 2 diabetes and frailty are improved when participating in the Band-Frail Program.

DETAILED DESCRIPTION:
Individuals considered fragile or frail and living with type 2 diabetes (T2D) have a 5-fold increased risk of being moved to a long-term care facility and a 4-fold increased risk of an emergency department visit. In 2013, the Mid-Frail study found that 16 weeks of combined exercise, diet, and education intervention significantly improved functional abilities in older adults living with T2D and frailty.

The goal of The Band-Frail Study is to implement an adapted version of the Mid-Frail program in New Brunswick (NB), while ensuring its sustainability by leveraging existing resources in the future as NB has one of the highest rates of diabetes in Canada and one of the highest average age of residents.

This project will include adults aged 65 years and above living with T2D and frailty across the province of New Brunswick (NB). Participants will meet in groups of 4-8 people twice a week for 16 weeks. One session will consist of diabetes management education delivered by a Certified Diabetes Educator and elastic band resistance training, while the second session will only involve the elastic band resistance training.

Participants will undergo pre- and post-testing including questionnaires, physical function tests, and interviews to assess the viability of this program in the province and determine the physical and psychological benefits.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years old
* Classified as frail or pre-frail on Fried's Frailty Scale
* Self-reported diagnosis of type 2 diabetes
* Not physically active (3+ days of physical activity per week)

Exclusion Criteria:

* Aged under 65 years old
* Classified as robust of Fried's Frailty Scale
* Not diagnosed with type 2 diabetes
* Regularly physically active (3+ days of physical activity per week)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Physical Functioning | 16 weeks
  Physical functioning will be measured using the Short Physical Performance Battery (SPPB). The SPPB is a three-part standardized test including balance, gait, and chair stand components each scored out of 4 points for a total possible score ranging from 0 to 12 points. A higher SPPB score suggests high levels of physical functioning, while a lower SPPB score suggests functional limitations.

SECONDARY OUTCOMES:
Frailty Status | 16 weeks
  Frailty status will be measured using Fried's Frailty Scale. The scale includes five frailty criteria: unintentional weight loss, exhaustion, low physical activity, slowness, and weak grip strength.
  Participants will be scored in each of the five criteria and then given a cumulative score ranging from 0 to 5 to represent their frailty status. Participants who score three or more criteria will be considered frail, individuals who score one or two criteria will be considered pre-frail, and those who score zero criteria will be considered robust (non-frail).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick- Faculty of Kinesiology, Fredericton, New Brunswick, Canada